CLINICAL TRIAL: NCT03427827
Title: Camrelizumab (PD-1 Antibody) Compared With Best Supportive Care After Chemoradiotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma: a Multi-center, Randomised Controlled, Phase 3 Trial (DIPPER)
Brief Title: PD-1 Antibody Versus Best Supportive Care After Chemoradiation in Locoregionally Advanced Nasopharyngeal Carcinoma
Acronym: DIPPER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-097-01
Record Dates: First submitted 2018-02-03; First posted 2018-02-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: PD-1 antibody; Adjuvant treatment; Immune checkpoint inhibitors
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant PD-1 antibody arm (Experimental): Patients randomized to this arm will receive PD-1 antibody (SHR-1210), 200mg, ivdrip (>30 minutes), d1, q3w × 12 cycles, begining at 4-6 weeks after chemoradiation
  Interventions: Drug: Camrelizumab
- Best supportive care (No Intervention): Patients randomized to this arm will receive best supportive care after chemoradiation

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab is an antibody targeting PD-1 developed by Jiangsu Hengrui Medicine, China.
  Other Names: SHR-1210
  Arms: Adjuvant PD-1 antibody arm

SUMMARY:
This trial is aimed to investigate whether adjuvant PD-1 antibody treatment could improve survival in locoregionally advanced nasopharyngeal carcinoma compared to best supportive care.

DETAILED DESCRIPTION:
In this multicenter, randomised controlled, phase 3 trial, patients with stage III-IVA (AJCC/UICC 8th system, except T3-4N0 and T3N1) non-metastatic nasopharyngeal carcinoma will be randomized in a 1:1 ratio to recieve PD-1 antibody for 12 doses every 3 weeks or best supportive care after curative chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed nasopharyngeal carcinoma.
* Tumor staged as III-IVA (AJCC 8th, except T3N0-1 or T4N0).
* Completed protocol-specified curative chemoradiotherapy, including gemcitabine and cisplatin induction chemotherapy, intensity-modulated radiotherapy, and concurrent cisplatin chemotherapy.
* Completion of the last radiation dose within 1 to 42 days before randomization
* Eastern Cooperative Oncology Group performance status ≤1.
* Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.
* Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.
* Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
* Patients must be informed of the investigational nature of this study and give written informed consent.
* Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug.

Exclusion Criteria:

* Age > 65 or < 18.
* Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA >1×10e3 copies/ml or 200IU/ml
* Hepatitis C virus (HCV) antibody positive
* Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
* Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroid will be allowed.
* Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB over 1 year ago will be allowed.
* Has a known history of interstitial lung disease.
* Has received a live vaccine within 30 days before informed consent or will receive a live vaccine in the near future.
* Is pregnant or breastfeeding.
* Prior malignancy within 5 years, except in situ cancer, adequately treated non-melanoma skin cancer, and papillary thyroid carcinoma.
* Has known allergy to large molecule protein products or any compound of camrelizumab.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
failure-free survival | 3 years
  calculated from the date of randomisation to the date of locoregional failure, distant failure, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
overall survival | 5 years
  calculated from date of randomisation to death
distant metastasis-free survival | 3 years
  calculated from date of randomisation to the first distant failure
locoregional recurrence-free survival | 3 years
  calculated from date of randomisation to the first locoregional failure
adverse events (AEs) and severe adverse events (SAE) | 3 years
  graded according to NCI CTCAE v5.0
quality of life (QoL) | 3 years
  the change of QoL from randomization to 36 months after chemoradiation, graded according to EORTC QLQ-C30 V3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD, Principal Investigator — Sun Yat-sen University
Locations (11):
- China (11):
  - First People's Hospital of Foshan, Foshan, Guangdong
  - Guangzhou Medical University Cancer Hospital, Guangzhou, Guangdong
  - Panyu central hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Tongji Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Xijing Hospital, Fourth Military Medical University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
Complete de-identified patient data set
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: For 2 years started from 12 months after publication of the primary trial report.
Access Criteria: Authoritative researchers who provide a methodologically sound proposal for individual participant data meta-analysis.

REFERENCES:
- [Derived] Liang YL, Liu X, Shen LF, Hu GY, Zou GR, Zhang N, Chen CB, Chen XZ, Zhu XD, Yuan YW, Yang KY, Jin F, Hu WH, Xie FY, Huang Y, Han F, Tang LL, Mao YP, Lu LX, Sun R, He YX, Zhou YY, Long GX, Tang J, Chen LS, Zong JF, Jin T, Li L, Lin J, Huang J, Gong XY, Zhou GQ, Chen L, Li WF, Chen YP, Xu C, Lin L, Huang SH, Huang SW, Wang YQ, Huang CL, Feng HX, Hou M, Chen CH, Zheng SF, Li YQ, Hong SB, Jie YS, Li H, Yun JP, Zang SB, Liu SR, Lin QG, Li HJ, Tian L, Liu LZ, Zhao HY, Li JB, Lin AH, Liu N, Zhang Y, Guo R, Ma J, Sun Y. Adjuvant PD-1 Blockade With Camrelizumab for Nasopharyngeal Carcinoma: The DIPPER Randomized Clinical Trial. JAMA. 2025 May 13;333(18):1589-1598. doi: 10.1001/jama.2025.1132. PMID 40079940
- [Derived] Huang SW, Jiang W, Xu S, Zhang Y, Du J, Wang YQ, Yang KY, Zhang N, Liu F, Zou GR, Jin F, Wu HJ, Zhou YY, Zhu XD, Chen NY, Xu C, Qiao H, Liu N, Sun Y, Ma J, Liang YL, Liu X. Systemic longitudinal immune profiling identifies proliferating Treg cells as predictors of immunotherapy benefit: biomarker analysis from the phase 3 CONTINUUM and DIPPER trials. Signal Transduct Target Ther. 2024 Oct 23;9(1):285. doi: 10.1038/s41392-024-01988-w. PMID 39438442